CLINICAL TRIAL: NCT01612520
Title: Telecoaching of People With Type 2 Diabetes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Irina Odnoletkova, PhD Student in Biomedical sciences, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S53665
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes Mellitus; Telenursing
Keywords: type 2 Diabetes Mellitus; telenursing; RCT; economic analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telecoaching (Active Comparator)
  Interventions: Behavioral: telecoaching
- control (No Intervention)

INTERVENTIONS:
Behavioral: telecoaching — The COACH program trains patients to 'drive' the process of achieving and maintaining the target levels for their risk factors while working in association with their GP. The telephone coaching is aimed at improving self-efficacy by adhering to the prescribed therapy and making relevant behavior changes.
  The coaching model is a continuous five-stage coaching cycle: Stage 1. Finding out what the patient knows; Stage 2. Telling the patient what they should know; Stage 3. Assertiveness training; Stage 4. Setting an action plan; Stage 5. Reassessment at the next coaching session (monitoring).
  The coach monitors and registers: the biomedical risk factors, the lifestyle/behavioral risk factors and use of the recommended medications. Coaching is focused on eliminating the knowledge gap and motivating the patient to apply the appropriate lifestyle and medical therapy.
  Arms: telecoaching

SUMMARY:
The objective of the study is to analyze the effectiveness and the cost-effectiveness of telecoching in improving glyceamic control and other modifiable risk factors in patients with type 2 diabetes compared to usual care only.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes between 18 and 75 years old on the day of the selection

Exclusion Criteria:

* Debilitating coexisting medical condition (e.g. dialysis, mental illness, cancer)
* Residents of long term care facilities
* Pregnancy
* Incapable of telephone communication in Dutch

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
the absolute change in HbA1c | baseline; 6 months and 18 months

REFERENCES:
- [Derived] Odnoletkova I, Buysse H, Nobels F, Goderis G, Aertgeerts B, Annemans L, Ramaekers D. Patient and provider acceptance of telecoaching in type 2 diabetes: a mixed-method study embedded in a randomised clinical trial. BMC Med Inform Decis Mak. 2016 Nov 9;16(1):142. doi: 10.1186/s12911-016-0383-3. PMID 27825340
- [Derived] Odnoletkova I, Ramaekers D, Nobels F, Goderis G, Aertgeerts B, Annemans L. Delivering Diabetes Education through Nurse-Led Telecoaching. Cost-Effectiveness Analysis. PLoS One. 2016 Oct 11;11(10):e0163997. doi: 10.1371/journal.pone.0163997. eCollection 2016. PMID 27727281
- [Derived] Odnoletkova I, Goderis G, Nobels F, Aertgeerts B, Annemans L, Ramaekers D. Nurse-led telecoaching of people with type 2 diabetes in primary care: rationale, design and baseline data of a randomized controlled trial. BMC Fam Pract. 2014 Feb 4;15:24. doi: 10.1186/1471-2296-15-24. PMID 24495633